CLINICAL TRIAL: NCT05183230
Title: WellPATH-PREVENT: A Mobile Intervention for Middle-Aged and Older Adults Hospitalized for Suicidal Ideation or Attempt
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-12024207; R61MH128516 (NIH); R33MH128516 (NIH)
Record Dates: First submitted 2021-12-20; First posted 2022-01-10 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Suicide, Attempted; Suicidal Ideation; Depression
Keywords: Older Adults; Middle Aged Adults
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The research assistants administering the assessments will be blind to participant randomization in the R33 phase.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Proof-of-Concept WellPATH-PREVENT (R61) (Experimental)
  Interventions: Behavioral: WellPATH-PREVENT
- Optimized WellPATH-PREVENT (R33) (Experimental)
  Interventions: Behavioral: Optimized WellPATH-PREVENT
- Attention Control Usual Care (R33) (No Intervention): The AC-UC group will parallel the delivery of the WellPATH-PREVENT intervention and will also include: a) meetings during hospitalization: a non-clinical member of the team will present the control tablet and explain its use; b) scheduled or requested meetings through zoom: to parallel the delivery of WellPATH-PREVENT. The tablet will still have a link to schedule a meeting with a non-clinician member of the team. The meetings will focus on issues that the patient may have in using the tablet. There will not be any therapeutic or psychological interaction between participants in the control group and the team. The experimental and the control group will also be under usual outpatient care, which is arranged during the hospitalization by the inpatient treatment team.

INTERVENTIONS:
Behavioral: WellPATH-PREVENT — WellPATH-PREVENT is a novel personalized, easy to use, mainly stand-alone mobile intervention which focuses on the exclusive use of the WellPATH tablet app and includes training meetings during hospitalization, and virtual post-discharge coaching meetings. The meetings aim to: a) identify stressors and triggers of negative emotions associated with increased suicidal ideation or with suicidal behavior; b) develop techniques (text or video) to increase cognitive reappraisal ability; c) incorporate the techniques into the WellPATH app and promote the use of WellPATH during stressful incidents, triggers of negative emotions, or scheduled brief training sessions; and d) remotely update the triggers, negative emotions, and techniques in the app.
  Arms: Proof-of-Concept WellPATH-PREVENT (R61)
Behavioral: Optimized WellPATH-PREVENT — The Optimized WellPATH-PREVENT intervention will be as described above, but based on the results of the Proof-of-Concept (R61) Phase, an expert committee will help select the duration (6 or 12 weeks) that shows greater improvement in cognitive reappraisal.
  Arms: Optimized WellPATH-PREVENT (R33)

SUMMARY:
The goal of this project is to test whether WellPATH-PREVENT (a novel, mobile psychosocial intervention) improves a specific aspect of emotion regulation, i.e., cognitive reappraisal ability, and reduces suicide risk in middle-aged and older adults (50-90 years old) who have been discharged after a suicide-related hospitalization (i.e. for suicidal ideation or suicide attempt).

DETAILED DESCRIPTION:
R61 Phase: In this "proof-of-concept" phase, interventionists will administer 12 weeks of WellPATH-PREVENT in 40 middle-aged and older adults who have been discharged after being hospitalized for suicidal ideation or suicide attempt. The interventionist will help the patient incorporate the appropriate data (i.e., triggers, negative emotions, cognitive reappraisal techniques) into the tablet, train the patients on how to use the tablet, and coach them during the 12 weeks. There will be 4 assessments: At study entry (admission/during hospitalization), hospital discharge, 6, and 12 weeks. An EEG will be conducted upon entry into the study, at Week 6, and at Week 12.

R33 Phase: 75 middle-aged and older adults who have been recently discharged after a hospitalization for suicidal ideation or attempt will be recruited and randomized to an optimized version of WellPATH-PREVENT (Week 6 and Week 12 duration based on R61 results) or to Attention Control-Usual Care with a tablet (AC-UC). There will be 5 assessments: At study entry (admission/during hospitalization), discharge, 6, 12 and 24 weeks. Participants who exit the study prior to completion will be invited to have an assessment before termination as close to the scheduled time point as possible. Psychiatrically re-hospitalized participants will not be dropped from the study but will have an additional assessment and will continue the assessments as scheduled based on their initial hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* 50-90 years old
* Diagnosis (based on a modified SCID-5 Clinical Trials Version to assess DSM-5 diagnoses): Any DSM-5 except: current diagnosis of Psychotic Disorder; diagnosis of Dementia
* Recent hospitalization for suicidal ideation or suicide attempt; at hospital admission, Columbia Suicide Severity Rating Scale (CSSR-S) ≥ 2, "Non-specific Active Suicidal Thoughts."
* We will also include patients on psychotropics and on after-care community psychotherapy.

Exclusion Criteria:

* Current diagnosis of Psychotic Disorders; Diagnosis of Dementia
* Cognitive Impairment (MMSE ≤ 24)
* Acute or severe medical illness (i.e., delirium; decompensated cardiac, liver or kidney failure; major surgery; stroke or myocardial infarction during the three months prior to entry
* Aphasia, sensory problems, and/or inability to speak English.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Event Related Potential - Late Positive Potential (ERP/LPP) - R61 | Study Entry, Week 6, Week 12
  ERP is used to measure the amplitude (magnitude) of electrocortical activity (measured in μV) during an emotion regulation task.
Change in Event Related Potential - Late Positive Potential (ERP/LPP) - R33 | Study Entry, Week 6, Week 12, Week 24
  ERP is used to measure the amplitude (magnitude) of electrocortical activity (measured in μV) during an emotion regulation task.
Change in Self-Reported Affect - R61 | Study Entry, Week 6, Week 12
  Self-reported affect is used to study changes in negative emotions during an EEG emotion regulation task. It is based on a participant's rating of negative emotions (Likert scale: 1-5; 5 most negative) during the task.
Change in Self-Reported Affect - R33 | Study Entry, Week 6, Week 12, Week 24
  Self-reported affect is used to study changes in negative emotions during an EEG emotion regulation task. It is based on a participant's rating of negative emotions (Likert scale: 1-5; 5 most negative) during the task.
Change in Emotion Regulation (Cognitive Reappraisal Subscale of ER Questionnaire) - R61 | Study Entry, Week 6, Week 12
  ERQ is an interviewer-administered instrument to evaluate cognitive reappraisal ability. Scores can range from 1-7, where higher scores indicate greater use of emotion regulation strategies and lower scores indicate less frequent use of such strategies.
Change in Emotion Regulation (Cognitive Reappraisal Subscale of ER Questionnaire) - R33 | Study Entry, Week 6, Week 12, Week 24
  ERQ is an interviewer-administered instrument to evaluate cognitive reappraisal ability. Scores can range from 1-7, where higher scores indicate greater use of emotion regulation strategies and lower scores indicate less frequent use of such strategies.
Change in Client Satisfaction with Treatment (CSQ) - R61 | Week 6, Week 12
  Client Satisfaction Questionnaire is a self-report that measures patient satisfaction with intervention/treatment. Scores can range from 3-12, where higher values indicate higher satisfaction.
Change in Client Satisfaction with Treatment (CSQ) - R33 | Week 6, Week 12, Week 24
  Client Satisfaction Questionnaire is a self-report that measures patient satisfaction with intervention/treatment. Scores can range from 3-12, where higher values indicate higher satisfaction.
Change in Suicide Risk - Columbia Suicide Severity Scale (C-SSRS) - R61 | Weekly from Study Entry to Week 12 (R61)
  C-SSRS is used to measure intensity of suicidal ideation. Scores range from 0-5, where higher scores indicate more severe ideation.
Change in Suicide Risk - Columbia Suicide Severity Scale (C-SSRS) - R33 | Weekly from Study Entry to Week 24
  C-SSRS is used to measure intensity of suicidal ideation. Scores range from 0-5, where higher scores indicate more severe ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Kiosses, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - New York Presbyterian Hospital/Weill Cornell Medicine, New York, New York
  - Weill Cornell Institute of Geriatric Psychiatry, Weill Cornell Medicine, White Plains, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from this study is submitted to the National Database for Clinical Trials related to Mental Illness (NDCT). The NDCT is run by NIH and allows researchers studying mental health to collect and share information with each other. Researchers must apply to NIH in order to be allowed access to the data for 1 year's time; after which they must re-apply.
Time Frame: Data will be available as per NIH's data sharing policy.
Access Criteria: Access criteria is determined by NIH and can be requested by applying online.
URL: http://nda.nih.gov/